CLINICAL TRIAL: NCT01881347
Title: Randomized Crossover Study of The Effects of Resveratrol on Endothelial Function in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effects of Resveratrol on Endothelial Function in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-32036; 5P01HL068758-10 (NIH)
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus
Keywords: endothelium; mitochondria; reactive oxygen species; vascular biology; arterial stiffness; nitric oxide
MeSH Terms: conditions — Diabetes Mellitus | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active First (Experimental): Active resveratrol first, placebo second
  Interventions: Dietary Supplement: Resveratrol; Dietary Supplement: Placebo
- Placebo first (Experimental): Placebo first, active resveratrol second
  Interventions: Dietary Supplement: Resveratrol; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Resveratrol 100 mg daily for 2 weeks followed by resveratrol 300 mg daily for 2 weeks.
Dietary Supplement: Placebo — Placebo 100 mg daily for 2 weeks followed by placebo 300 mg daily for 2 weeks.

SUMMARY:
The present study is designed to test the hypothesis that resveratrol supplementation will improve the function of the endothelium in patients with type 2 diabetes mellitus.

The function of the endothelium will be tested with a non-invasive technique that uses ultrasound to measure the amount of dilation that occurs in the brachial artery following 5-minute cuff occlusion. To help us understand potential mechanisms of benefit, we will also collect blood, urine, and cell samples and test the effects of treatment on protein expression, nitric oxide production, and function of mitochondria.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age over 21 years old
* Body mass index less than 38 kg/m2
* Clinical stable type 2 diabetes mellitus

Exclusion Criteria:

* Women who are lactating or pregnant
* Treatment with an investigations product within 30 days of screening
* Clinically evident major illness of other organ systems, including cancer, renal failure, or other conditions in the opinion of the investigators that would make clinical study inappropriate
* Liver transaminase levels greater than 3 times the upper limit of normal
* History of psychological illness or condition that would interfere with the subject's ability to understand the requirements of the study
* Vitamin supplements exceeding two times the recommended daily allowance
* Resveratrol or other dietary supplements except for a daily multivitamin

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Brachial artery flow mediated dilation | 2 hours, 2 weeks, and 4 weeks

SECONDARY OUTCOMES:
Change from Baseline in Fingertip peripheral arterial tonometry | 2 hours, 2 weeks, and 4 weeks
Change from Baseline in Carotid femoral pulse wave velocity | 4 weeks
Change from Baseline in Reactive hyperemia | 2 hours, 2 weeks, 4 weeks

OTHER OUTCOMES:
Change from Baseline in Serum glucose | 2 and 4 weeks
Change from Baseline in Serum insulin | 2 and 4 weeks
Change from Baseline in Mononuclear cell mitochondrial DNA damage | 4 weejs
Change from Baseline in Mononuclear cell mitochondrial mass | 4 weeks
Change from Baseline in Mononuclear cell mitochondrial production of reactive oxygen species | 4 weeks
Change from Baseline in Endothelial cell gene expression | 4 weeks
Change from Baseline in Endothelial cell protein expression | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hamburg, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No